CLINICAL TRIAL: NCT00204854
Title: Telephone and Mail Intervention for Alcohol Use Disorders
Acronym: TAMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1999-514; 1R01AA012826 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-01

CONDITIONS: Alcohol Use Disorders
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: telephone counseling

SUMMARY:
Randomized controlled trial and benefit-cost study of a telephone and mail intervention for non-treatment-seeking primary care patients with alcohol abuse or dependence

ELIGIBILITY:
Inclusion Criteria:

* primary care patients with DSM-IV alcohol abuse or dependence

Exclusion Criteria:

* pregnancy
* suicidality
* alcohol treatment in prior 3 months

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900
Dates: Start 2001-12; Primary Completion 2004-06 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Self-reported alcohol consumption in the prior 28 days
Number of risky drinking days in the prior 28 days

SECONDARY OUTCOMES:
Health care utilization
car crashes
criminal justice system involvement

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Brown, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States